CLINICAL TRIAL: NCT01380535
Title: A Randomized Controlled Study of Extracorporeal Photopheresis (ECP) Therapy With UVADEX for the Treatment of Patients With Moderate to Severe Chronic Graft-versus-Host Disease (cGvHD)
Brief Title: Extracorporeal Photopheresis (ECP) With Methoxsalen for Chronic Graft Versus Host Disease (cGVHD)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-005; 2010-022780-35 (EudraCT Number)
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: Extracorporeal photopheresis therapy; Methoxsalen; cGVHD; hematopoietic stem cell transplantation
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Methoxsalen; Photopheresis; Standard of Care

STUDY DESIGN:
Intervention Model Description: Pilot Study for the 2015 NIH Consensus Criteria to inform the design of subsequent studies
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ECP Methoxsalen + Standard of Care (Experimental): Participants receive methoxsalen administered via ECP in addition to standard of care
  Interventions: Drug: ECP Methoxsalen; Drug: Standard of Care
- Standard of Care (Active Comparator): Participants receive standard of care only
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: ECP Methoxsalen — Methoxsalen delivered by ECP
  Other Names: Uvadex; Extracorporeal photopheresis (ECP)
  Arms: ECP Methoxsalen + Standard of Care
Drug: Standard of Care — Tapered prednisone with cyclosporine or tacrolimus via oral administration, consistent with local institutional practice (corticosteroids and cyclosporine A/tacrolimus)
  Other Names: Reference therapy

SUMMARY:
Chronic graft-versus-host disease (cGVHD) is a long-lasting complication that can occur after transplants. The transplanted cells seem to fight with the patient's own cells.

Extracorporeal photopheresis (ECP) is a fairly new procedure for cGVHD. The participant gets a port to hook up to a machine. The machine removes the white blood cells, mixes them with a light-sensitive drug, shines light on it, and puts all the blood back in.

This study will find out if patients respond better if they get ECP with methoxsalen, in addition to the pills normally used to treat cGVHD.

DETAILED DESCRIPTION:
The investigation of extracorporeal photopheresis (ECP) plus standard of care (SoC) (SoC+ECP) in chronic graft-versus-host disease (cGVHD) within prospective, randomized clinical studies is limited, despite its frequent clinical use.

This phase 1/pilot study was the first randomized, prospective study to investigate ECP use as first-line therapy in cGVHD, based on the 2015 National Institutes of Health (NIH) consensus criteria for diagnosis and response assessment.

Adult patients with new-onset (≤3 years of hematopoietic stem cell transplantation) moderate or severe cGVHD were randomized 1:1 to 26 weeks of SoC+ECP vs SoC (corticosteroids and cyclosporine A/tacrolimus) between 2011 and 2015. The primary endpoint was overall response rate (ORR), defined as complete or partial response, at week 28 in the intention-to-treat population (ITT).

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion in this trial, the patient must have moderate to severe chronic graft-versus-host disease [defined by the National Institutes of Health (NIH) 2015 Consensus Criteria] that started within 3 years after hematopoietic stem cell transplantation (HSCT).

Exclusion Criteria:

* Is intolerant to corticosteroids or hypersensitive to methoxsalen
* Received certain treatments during time periods disallowed by protocol
* Has infections and/or requires treatment that (per protocol or in the opinion of the investigator) might compromise:

  1. safety and well-being of participant or offspring
  2. safety of study staff
  3. analysis of results

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (32):
- United States (11):
  - University of Miami Hospital, Miami, Florida
  - Indiana Blood and Marrow Transplantation Research, Indianapolis, Indiana
  - Tulane University Health Sciences Center, 1430 Tulane Avenue, Rm 7551,, New Orleans, Louisiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York Presbyterian Hospital, New York, New York
  - Stony brook university medical Center, Stony Brook, New York
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Medical City Dallas Hospital,Transplant center, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Methodist healthcare system of san Antonio, San Antonio, Texas
- General Hospital of Vienna (Medical University of Vienna), Vienna, Austria
- France (3):
  - Hopital Saint Antoine, Saint-Antoine, Paris
  - CHU de Nantes, Nantes
  - Hospital Saint Louis, Paris
- Germany (9):
  - Universitätsklinik Köln, Cologne
  - Universitäts-Klinikum Carl Gustav Carus, Dresden
  - Universitatsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Universitatskrankenhaus Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Universitätklinikum Mannheim, Mannheim
  - Medizinische Universitatsklinik, München
  - Uniklinik für Kinder und Jugendmedizin, Tübingen
- Egyesített Szent István és Szent László Kórház, Gyáli út 5-7,, Budapest, Hungary
- Italy (2):
  - A.O.U. Policlinico- Vittorio Emanuele, Catania
  - Universita de Genova - Ospedale S. Martino, Genova
- Spain (2):
  - Hospital Marques de Valdecilla, Santander, Cantabria
  - Santa Creu I Sant Pau, Barcelona
- United Kingdom (3):
  - Kings College Hospital, London, Greater London
  - University of Birmingham: Queen Elizabeth Hospital, Birmingham
  - Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jagasia M, Scheid C, Socie G, Ayuk FA, Tischer J, Donato ML, Batai A, Chen H, Chen SC, Chin T, Boodee H, Mitri G, Greinix HT. Randomized controlled study of ECP with methoxsalen as first-line treatment of patients with moderate to severe cGVHD. Blood Adv. 2019 Jul 23;3(14):2218-2229. doi: 10.1182/bloodadvances.2019000145. PMID 31332045
- See also: Cited article made available by the US National Library of Medicine, National Institutes of Health — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6650730/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in Austria, France, Germany, Italy, Hungary, Spain, the United Kingdom, and the United States. Enrollment started in November 2011, and the last patient visit occurred in March 2015.
Pre-assignment Details: All participants enrolled were included in the safety analysis set
Groups:
- ECP Methoxsalen + SoC: Participants receive ECP methoxsalen in addition to standard of care
- Standard of Care (SoC): Participants receive only standard of care
Period: Overall Study
Arm/Group | ECP Methoxsalen + SoC | Standard of Care (SoC)
Started | 29 | 31
Baseline Population (All enrolled participants) | 29 | 31
Safety Population (All randomized participants who received at least 1 dose of study treatment, per treatment received.) | 28 | 28
Intent-to-treat Population (All randomized subjects with baseline and post-treatment measurements, per assigned treatment) | 29 | 24
Completed | 22 | 16
Not Completed | 7 | 15
Not completed — Adverse Event | 3 | 3
Not completed — Death | 3 | 0
Not completed — Study site closed | 0 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Lack of Efficacy | 0 | 3

BASELINE CHARACTERISTICS:
Population: All participants enrolled and included in the safety analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | ECP Methoxsalen + SoC | Standard of Care (SOC) | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 8 | 10 | 18
  45-64 years | 19 | 19 | 38
  65 years and over | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 22 | 18 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 3 | 5 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 24 | 46
  Black | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Other | 1 | 1 | 2
  Not Collected | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  Austria | 3 | 3 | 6
  Hungary | 4 | 4 | 8
  United States | 6 | 6 | 12
  Italy | 0 | 3 | 3
  United Kingdom | 1 | 1 | 2
  France | 4 | 6 | 10
  Germany | 11 | 7 | 18
  Spain | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Overall Response at Week 28
Description: Participants with overall response included those with partial response or complete response, according to study staff who did not know which treatment they received (blinded assessment).
Time Frame: Week 28
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ECP Methoxsalen + SoC | Standard of Care (SoC)
Number analyzed (Participants) | 29 | 24
Participants | 20 | 14
Statistical Analysis 1: Comparison: ECP Methoxsalen + SoC vs Standard of Care (SoC); Test type: Other; p = 0.373, Fisher Exact

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were recorded from the start of treatment through Week 28.
Description: Treatment emergent adverse events (TEAEs) are unpleasant events not there before the medical treatment, or that were there, but got worse or happened more often after the treatment. Both serious and non-serious adverse events reported here are TEAEs. All-cause mortality is based on baseline population, while serious adverse events and non-serious adverse events are based on the safety population.
Arm/Group | ECP Methoxsalen + SoC | Standard of Care (SoC)
All-Cause Mortality (participants affected / at risk) | 4/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 8/28 | 9/28
Other Adverse Events (participants affected / at risk) | 26/28 | 24/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ECP Methoxsalen + SoC (N=28) | Standard of Care (SoC) (N=28)
Cardiac Failure (Cardiac disorders) | 0 | 1
Thyroiditis subacute (Endocrine disorders) | 1 | 0
Graft versus host disease in liver (Immune system disorders) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 0 | 1
Toxoplasmosis (Infections and infestations) | 1 | 0
Viraemia (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 2
Polyneuropathy (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ECP Methoxsalen + SoC (N=28) | Standard of Care (SoC) (N=28)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4
Dry Eye (Eye disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Asthenia (General disorders) | 1 | 2
Fatigue (General disorders) | 5 | 1
Oedema peripheral (General disorders) | 2 | 4
Pyrexia (General disorders) | 0 | 4
Epstein-Barr virus infection (Infections and infestations) | 1 | 3
Rhinitis (Infections and infestations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 2
Blood cholesterol increased (Investigations) | 3 | 1
Blood creatinine increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 2
Blood pressure increased (Investigations) | 1 | 3
Blood urea increased (Investigations) | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 4 | 3
Platelet count decreased (Investigations) | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4
Myopathy (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 2 | 3
Sleep disorder (Psychiatric disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 2
Hypertension (Vascular disorders) | 9 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Paraesthesia (Nervous system disorders) | 2 | 2
Dizziness (Nervous system disorders) | 4 | 2
Tremor (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 2 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2

LIMITATIONS AND CAVEATS:
Long term follow-up (LTFU) safety data were provided to health authorities in safety reports; not the 28-week protocol.

LTFU pre-specified outcome measures previously entered in error were removed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less